CLINICAL TRIAL: NCT00100997
Title: A Phase 1, Multicenter, Open-Label, Dose-Escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of Intravenously Administered CNF1010 )17-(Allylamino)-17-Demethoxygeldanamycin [17-AAG]) in Patients With Gleevec-Resistent Chronic Myelogenous Leukemia
Brief Title: 17-N-Allylamino-17-Demethoxygeldanamycin in Treating Patients With Chronic Phase Chronic Myelogenous Leukemia That Did Not Respond to Imatinib Mesylate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: UCLA-0408048-01; CDR0000407499 (Registry Identifier: PDQ (Physician Data Query)); CTC-CNF1010; CTC-CNF1010-CML-04001
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2005-05

CONDITIONS: Leukemia
Keywords: chronic myelogenous leukemia, BCR-ABL1 positive; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — tanespimycin

INTERVENTIONS:
Drug: tanespimycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as 17-N-allylamino-17-demethoxygeldanamycin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. It may also stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of 17-N-allylamino-17-demethoxygeldanamycin in treating patients with chronic phase chronic myelogenous leukemia that did not respond to imatinib mesylate.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and dose-limiting toxicity of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG), in terms of frequency, severity, and duration of treatment-emergent adverse events, in patients with imatinib mesylate-resistant Philadelphia chromosome (Ph)-positive chronic phase chronic myelogenous leukemia.
* Determine the pharmacokinetics of this drug and its primary metabolite (17-amino-17-demethoxygeldanamycin) in these patients.

Secondary

* Determine the hematologic response rate, in terms of WBC count, platelet count, and assessment of blast cells in peripheral blood, in patients treated with this drug.
* Determine the cytogenic response rate, in terms of Ph-positive progenitor cells in the bone marrow, in patients treated with this drug.
* Assess the effect of this drug on pharmacodynamic markers (i.e., CRKL phosphorylation, BCR-ABL kinase activity, and BCR-ABL, RAF kinase, and HSP70 expression) in these patients.

OUTLINE: This is an open label, dose-escalation, multicenter study.

Patients receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) IV over 15 minutes or 1 hour (depending on the dose administered) once on days 1, 4, 8, 11, 15, 18, 22, and 25. Treatment repeats every 28 days for up to 3 courses in the absence of unacceptable toxicity or disease progression. Eligible patients may receive additional courses of 17-AAG at the discretion of the investigator.

Cohorts of 3-6 patients receive escalating doses of 17-AAG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 10 additional patients are treated at the MTD.

Patients are followed for 1 month.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic phase chronic myelogenous leukemia

  * Philadelphia chromosome (Ph)-positive disease
* Hematologic resistence after treatment with imatinib mesylate (400 mg per day or maximum tolerated dose [MTD]) as defined by 1 of the following criteria:

  * Loss of complete hematologic response, defined as WBC count OR platelet count > upper limit of normal (ULN) on 2 separate occasions at least 2 weeks apart that cannot be attributed to other etiologies
  * Absolute increase of ≥ 30% in Ph-positive cells while on a stable dose of imatinib mesylate for at least 6 months* NOTE: *Patients meeting this criterion are not eligible for enrollment into the expanded MTD cohort
* Less than 15% blasts in peripheral blood or bone marrow AND < 30% blasts and promyelocytes in peripheral blood or bone marrow

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin < 1.5 times ULN (3 mg/dL for patients with Gilbert's syndrome)
* ALT or AST < 2 times ULN
* No known hepatitis positivity

Renal

* Creatinine < 1.5 times ULN OR
* Creatinine clearance > 60 mL/min

Cardiovascular

* No New York Heart Association class III or IV cardiac disease

Pulmonary

* No severe debilitating pulmonary disease, including any of the following:

  * Dyspnea at rest
  * Significant shortness of breath
  * Chronic obstructive pulmonary disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after study participation
* No known HIV positivity
* No psychological or social condition that would preclude study compliance
* No addictive disorder that would preclude study compliance
* No family problems that would preclude study compliance
* No known allergy or sensitivity to soy or other excipient components of study drug
* No other illness or condition that may affect safety of study treatment or evaluation of study endpoints

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 2 weeks since prior interferon
* No concurrent interferon

Chemotherapy

* More than 2 weeks since prior cytarabine (4 weeks for doses > 100 mg)
* More than 6 weeks since prior busulfan
* No concurrent cytarabine
* No concurrent hydroxyurea during the second study treatment course and beyond
* No concurrent anagrelide during the second study treatment course and beyond

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 2 days since prior imatinib mesylate
* More than 1 week since prior and no concurrent drugs that alter metabolism by cytochrome P450 3A4, including the following:

  * Diltiazem
  * Nifedipine
  * Verapamil
  * Fluconazole
  * Itraconazole
  * Ketoconazole
  * Lovastatin
  * Simvastatin
  * Indinavir
  * Nelfinavir
  * Ritonavir
  * Alprazolam
  * Diazepam
  * Midazolam
  * Triazolam
  * Phenobarbital
  * Phenytoin
  * Carbamazepine
  * Azithromycin
  * Clarithromycin
  * Erythromycin
  * Rifampin
  * Rifamycin
  * Astemizole
  * Terfenidine
  * Amiodarone
  * Cimetidine
  * Cisapride
  * Cyclosporine
  * Grapefruit juice
  * Hypericum perforatum (St. John's wort)
  * Warfarin
* More than 4 weeks since prior investigational drugs and recovered
* No concurrent imatinib mesylate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-10; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Sawyers, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States